CLINICAL TRIAL: NCT02085681
Title: Effectiveness of Tele-medicine in Identifying Diabetic Retinopathy Cases Attending Diabetologists' Clinics Compared to the Conventional Referral System
Brief Title: Study of Effectiveness of Telemedicine in Identifying Diabetic Retinopathy Cases
Acronym: DRTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aravind Eye Care System (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Sanil Joseph, Faculty, Aravind Eye Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WT097685MA
Record Dates: First submitted 2014-02-05; First posted 2014-03-13 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Screening; Tele-medicine; Retinal Imaging; Remote diagnosis
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tele-medicine (Experimental): Tele-medicine aided retinal imaging and referral to eye hospital
  Interventions: Other: Tele-medicine
- Conventional Referral (Other): Patients will be counselled on the importance of eye examination and will be referred to the eye hospital in the conventional manner.
  Interventions: Other: Conventional referral

INTERVENTIONS:
Other: Tele-medicine — Patients at the diabetes clinics will be subjected to non-mydriatic retinal imaging and the images will be transferred to the eye hospital via internet using a specified software - Aravind Diabetic Retinopathy Evaluation Software (ADRES) that enables a retinal specialist to read and grad the image and send the feedback immediately to the diabetes clinic. Based on the presence or absence of DR the patients will be referred to the eye hospital for detailed retinal examination.
  Other Names: Tele-medicine aided retinal imaging
  Arms: Tele-medicine
Other: Conventional referral — All eligible patients in the conventional arm will be counselled on the importance of eye screening and will be referred to the eye hospital
  Arms: Conventional Referral

SUMMARY:
The aim of this study is to compare the effectiveness of identifying diabetic retinopathy using tele-medicine based Digital Retinal Imaging in Diabetes Clinics with that of the conventional referral system.

Hypothesis: Tele-medicine based digital retinal imaging involving a diabetes centre will identify proportionately more diabetic patients with DR and lead to higher acceptance rate with subsequent ophthalmic referral and management

DETAILED DESCRIPTION:
The design is a cluster randomized trial of tele-medicine versus usual care in diabetic patients. The primary outcome of the study is the proportion of patients with confirmed DR at Aravind Eye Hospital (AEH). DR will be graded using the International Clinical Diabetic Retinopathy Disease Severity Scale. A sample size of 616 patients in both arms is required to detect a risk ratio of 1.8 or above at 90% power, 1% alpha and a design effect of 2. Eight clinics will be recruited and equally randomized to tele-medicine or usual care stratified by distance from AEH. Inclusion criteria include a confirmed diagnosis of diabetes, age over 50, no retinal exam in the previous year. In the tele-medicine arm patients will be offered fundus imaging and patients diagnosed with DR or probable DR will be counselled to visit AEH to confirm DR. In the usual care arm, the eligible patients will be counselled and referred to undergo an eye examination at AEH. In both the arms the counselling and the awareness creation materials will be standardized. Fundus imaging will be offered at the end of the study to those who refuse initially and all those in the usual arm who did not attend AEH.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients (as per ICD-9 code 250) in the age group of ≥50 years

Exclusion Criteria:

* Patients <50 years of age
* Already enrolled as study patients at the diabetes centre
* Patients screened for DR in free camps organized by the diabetes centre
* Diabetic patients who underwent retinal examination in the previous year prior to this intervention
* Patients with disability (physical or mental) who have difficulty in travelling to the eye hospital

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with confirmed Diabetic Retinopathy (DR) diagnosed at the eye hospital | 6 months
  Out of the patients referred from the diabetes clinics to the eye hospital, the number of patients with confirmed DR will be measured. This proportion will be compared between the two arms.

SECONDARY OUTCOMES:
The severity of diabetic retinopathy (DR) | 6 months
  Among patients confirmed with DR, the severity of the disease will be measured using standard classification (Diabetic Retinopathy Disease Severity Scale) approved by the American Academy of Ophthalmology
The acceptance rate for referral in each arm | 6 months
  Out of the patients referred from the diabetes clinic, the number of patients actually reported to the eye hospital will be measured.
Proportion of patients eligible for referral who had DR and who did not attend | 6 months
  Patients who are referred by not attended to the eye hospital will be followed up and examined to find out what proportion of them actually as DR

OTHER OUTCOMES:
Barriers to compliance | 6 months
  Patients will be interviewed to identify the barriers to compliance following the referral
Drivers of acceptance | 6 months
  Patients will be interviewed to identify the factors that encouraged them to visit the eye hospital following referral

CONTACTS AND LOCATIONS:
Overall Officials: Sanil Joseph, MHA, MSc, Principal Investigator — Lions Aravind Institute of Community Ophthalmology, Aravind Eye Hospital, Madurai, India; Ramasamy Kim, DO, DNB, Study Chair — Aravind Eye Hospital, Madruai, India; Thulasiraj Ravilla, MBA, Study Chair — Lions Aravind Institute of Community Ophthalmology, Aravind Eye Hospital, Madurai; Astrid Fletcher, MSc, PhD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India

REFERENCES:
- [Derived] Joseph S, Kim R, Ravindran RD, Fletcher AE, Ravilla TD. Effectiveness of Teleretinal Imaging-Based Hospital Referral Compared With Universal Referral in Identifying Diabetic Retinopathy: A Cluster Randomized Clinical Trial. JAMA Ophthalmol. 2019 Jul 1;137(7):786-792. doi: 10.1001/jamaophthalmol.2019.1070. PMID 31070699